CLINICAL TRIAL: NCT02509663
Title: Medico-economic Evaluation of the Balloon Sinuplasty as Mini-invasive Treatment of Frontal Sinusitis by a Randomized Multicenter Prospective Trial
Brief Title: Treatment of Chronic Frontal Sinusitis by a Simple Technique Using Dilation Balloons
Acronym: SIBA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the manufacturer of the device has been bought and the new company does not want to continue the study anymore
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 6190
Record Dates: First submitted 2015-07-17; First posted 2015-07-28 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Frontal Sinusitis
MeSH Terms: conditions — Frontal Sinusitis | interventions — Endoscopes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sinuplasty balloon (Active Comparator): Patients will receive the innovative health technology to treat frontal sinusitis : a balloon sinuplasty
  Interventions: Procedure: Functional Endoscopic Sinus Surgery; Device: Sinuplasty balloon
- Conventional surgical procedure (Active Comparator): Patients will be treated with the conventional procedure : a sinus surgery with rigide instrumentation
  Interventions: Procedure: Functional Endoscopic Sinus Surgery using rigide instrumentation; Device: Endoscope

INTERVENTIONS:
Procedure: Functional Endoscopic Sinus Surgery — Balloon Sinuplasty uses a small, flexible, balloon catheter to open up blocked sinus passageways and facilitate drainage of the mucus that builds up in patients suffering from frontal sinusitis symptoms. When the sinus balloon is inflated, it restructures and widens the walls of the sinus passageway while maintaining the integrity of the sinus lining.
  Arms: Sinuplasty balloon
Procedure: Functional Endoscopic Sinus Surgery using rigide instrumentation — FESS (Functional Endoscopic Sinus Surgery) using rigide instrumentation is conventional therapeutic strategy.
  The procedure works by cutting to remove bone and tissue to enlarge the sinus opening.
  Arms: Conventional surgical procedure
Device: Sinuplasty balloon — Balloon Sinuplasty uses a small, flexible, balloon catheter to open up blocked sinus passageways and facilitate drainage of the mucus that builds up in patients suffering from frontal sinusitis symptoms. When the sinus balloon is inflated, it restructures and widens the walls of the sinus passageway while maintaining the integrity of the sinus lining.
  Arms: Sinuplasty balloon
Device: Endoscope — FESS (Functional Endoscopic Sinus Surgery) using rigide instrumentation is conventional therapeutic strategy.
  The procedure works by cutting to remove bone and tissue to enlarge the sinus opening.
  Arms: Conventional surgical procedure

SUMMARY:
The sinuplasty balloon offers a more physiological first of the sinuses which minimizes risks associated to traditional surgery. Its atraumatic characteristic also helps to reduce the risk of bleeding (so any use of Pack), limit scarring ransom, reduce the post-operative pain, ensure faster return to daily life activities (reduction of the average length of hospitalization). Patient's quality of life would be improved (SNOT-22 questionnaire) and reduction of post-operative pain score seams decrease on EVA.

The economic impact of the sinuplasty balloon appears very favourable and fits into the strategy of development of the ambulatory practice.

DETAILED DESCRIPTION:
The primary objective is to estimate the cost-utility ratio of the sinuplasty balloon after frontal sinus surgery, compared to surgery by rigid instrumentation, in a randomized single-blind controlled study.

The secondary objectives is to compare:

* the two types of surgery
* the quality of life
* the feeling of pain in patients but also the occurrence of surgical times or complications between the two proposed techniques.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman of age ≥ to 18 years.
* Patient for which a frontal sinus surgery (Draf 1 type) is programmed for any type of frontal sinusitis unresponsive to drug treatment properly leads.
* Patient affiliated to a social protection scheme Written informed consent of the patient
* Signed informed consent

Exclusion Criteria:

* Polyposis sinonasal or other sinus to be the subject of a simultaneous complementary intervention
* Sinuso-nasal tumors
* Osteogenesis
* Fragile patients or patient needing gesture contraindicating surgery by rigid instrumentation
* Contraindication with balloon using
* Contraindication to general anesthesia
* Immunosuppressive therapy
* Patient under judicial protection
* Pregnancy or Breastfeeding
* Exclusion period determinated with concurrent participation in other experimental studies
* Contrast medium allergy background
* Impossibility to give the informed study documentation to the subject (emergency situation, lack of understanding, etc...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Cost-utility ratio | This ratio will be assessed for 12 months post surgery
  Cost-utility ratio will be assessed with :
  * cost difference between sinuplasty balloon and conventional surgery
  * utility difference of these two surgery procedures estimated with EQ-5D questionnaire outcomes

SECONDARY OUTCOMES:
Quality of the patient's life | This secondary outcome will be assessed for 12 month : at inclusion and at 1 Week , 3 weeks , 3 -6 and 12 months post surgery
  Patient's quality of life include the following exams :
  * EuroQoL EQ-5D Questionnaire
  * SNOT-22 questionnaire
Risks associated with intervention | This secondary outcome will be assessed for 12 month
  Risks associated with intervention include the following criteria :
  * Occurrence of surgical times
  * Occurrence of complications
  * Presence of opacification in the visible sinus CT
Economic impact of the sinuplasty balloon | economic impact of this inovative technique will be assessed from sinus intervention to month 12 post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Christian Debry, Principal Investigator — Strasbourg's University Hospitals
Locations (8):
- France (8):
  - Service ORL et de Chirurgie Cervico-Faciale Hôpital Pellegrin, Bordeaux
  - Service ORL, stomatologie et de Chirurgie Cervico-Faciale Centre Hospitalier Intercommunal de Créteil, Créteil
  - Service ORL et de Chirurgie Cervico-Faciale, Nantes
  - Service ORL et de Chirurgie Maxillo-Faciale et Plastique Hôpital Lariboisière, Paris
  - Service ORL Institut Arthur Vernes, Paris
  - Service ORL, chirurgie maxillo-faciale et audiophonologie CHU - Hôpital de la Miletrie, Poitiers
  - ORL and facial surgery department, Hautepierre Hospital, Strasbourg's University Hospitals, Strasbourg
  - Service ORL et de Chirurgie Cervico-Faciale Hôpital Larrey, Toulouse